CLINICAL TRIAL: NCT03478436
Title: Pharmacokinetics of DFD-09 (Doxycycline) Capsules, 40 mg in Skin of Healthy Volunteers Under Fed and Fasting Conditions - an Exploratory Microdialysis Study
Brief Title: Pharmacokinetics of Doxycycline in Skin of Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Collaborators: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Principal Investigator, Markus Zeitlinger, Assoc. Prof. Priv.-Doz. Dr., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Version 1.0 / 04.05.2016
Record Dates: First submitted 2018-03-08; First posted 2018-03-27 (Actual); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Rosacea
Keywords: pharmacokinetics; microdialysis; healthy volunteers
MeSH Terms: conditions — Rosacea | interventions — Doxycycline

STUDY DESIGN:
Intervention Model Description: parallel groups to compare outcomes between fed and fasting conditions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fed group (Other): 14 once daily oral doses of doxycycline 40 mg, preceded by a standardized high-fat, high-calorie breakfast
  Interventions: Drug: Doxycycline
- fasting group (Other): 14 once daily oral doses of doxycycline 40 mg in fasting conditions (no food allowed 8 hours prior to dosing)
  Interventions: Drug: Doxycycline

INTERVENTIONS:
Drug: Doxycycline — Doxycycline 40 mg capsules

SUMMARY:
This study explored the impact of food on skin and plasma pharmacokinetics of doxycycline

DETAILED DESCRIPTION:
Sub-antimicrobial dose doxycycline is approved for the treatment of rosacea. This work investigated the pharmacokinetics of doxycycline in skin and plasma of fed and fasting healthy volunteers receiving a 14-day treatment course with once daily 40 mg doxycycline. Dermal measurements were performed by means of in vivo microdialysis.

ELIGIBILITY:
Inclusion Criteria:

Healthy males

* Healthy, according to the medical history, ECG, vital signs, laboratory results and physical examination as determined by the Investigator/Sub-Investigator
* Signed written informed consent prior to inclusion in the study
* 18-45 years old inclusive
* BMI: 18.5 to 30 kg/m2
* SBP: 100-139 mmHg
* DBP: 55-89 mmHg
* PR: 55-100 bpm (measured after 5 min of rest, sitting position)
* ability to comprehend the full nature and purpose of the study, including possible risks and side effects
* ability to co-operate with the Investigator and to comply with the requirements of the entire study
* availability to volunteer for the entire study duration and willing to adhere to all protocol requirements

Exclusion Criteria:

Any clinically relevant abnormalities in ECG (12 leads)

* Any clinically relevant abnormal physical findings
* Any clinically relevant abnormal laboratory values indicative of physical illness
* Ascertained or presumptive hypersensitivity to the active principle and/or formulations ingredients of the study drug or to tetracyclines in general
* History of anaphylaxis to drugs or allergic reactions in general, which the Investigator considers may affect the outcome of the study
* Relevant history of malignancy, of renal, hepatic, cardiovascular, respiratory, gastrointestinal, musculoskeletal, skin, haematological, endocrine or neurological diseases that may interfere with the aim of the study
* Any psychiatric illnesses
* Presence of any skin condition that would interfere with the placement of microdialysis probes
* Any dermatological drug therapy on the surface of both thighs within 14 days before study day 1 of this study
* Use of any medication(including OTC) within 1 week prior to study day 1
* Use of any enzyme-modifying drugs, including strong inhibitors of cytochrome P450 (CYP) enzymes (such as cimetidine, fluoxetine, quinidine, erythromycin, ciprofloxacin, fluconazole, ketoconazole, diltiazem and HIV antivirals) and strong inducers of CYP enzymes (such as barbiturates, carbamazepine, glucocorticoids, phenytoin, rifampin and St John's Wort) within 1 month prior to study day 1
* Participation in another clinical study investigating another IMP within 1 month prior to study day 1
* Blood donations within 1 month prior to study day 1 or planned within 1 month after the last study-related blood draw
* History of drug or alcohol abuse (>2 drinks/day, defined according to USDA Dietary Guidelines 2005)
* other objections to study participation in the opinion of the Investigator

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2016-10-25 (Actual); Study Completion 2016-10-25 (Actual)

PRIMARY OUTCOMES:
AUC0-t | at day 14
  mg∙h/L

CONTACTS AND LOCATIONS:
Overall Officials: Markus Zeitlinger, Principal Investigator — Department of Clinical Pharmacology, Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No
publication in peer-reviewed journal